CLINICAL TRIAL: NCT02302157
Title: A Phase 1/2a Dose Escalation Study of AST-OPC1 in Subjects With Subacute Cervical Spinal Cord Injury
Brief Title: Dose Escalation Study of AST-OPC1 in Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lineage Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST-OPC1-01
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Cervical Spinal Cord Injury; Spine Injury; Spinal Cord Trauma
Keywords: Cervical spinal cord injury; AST-OPC1; SCiStar; OPC1; Neural cell; Trauma spinal cord; stemcell transplant; Cervical spine injury; Paralysis; Quadriplegia; Tetraplegia; Spine injury; oligodendrocyte progenitor cell; Subacute spinal cord injury
MeSH Terms: conditions — Spinal Injuries; Spinal Cord Injuries; Paralysis; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AST-OPC1 (Experimental): Open label, dose escalation, cross-sequential cohort of subjects who receive an injection or two injections of AST-OPC1 at a single time-point
  Interventions: Biological: AST-OPC1

INTERVENTIONS:
Biological: AST-OPC1 — One injection of 2 million or 10 million AST-OPC1 cells, or 2 injections of 10 million AST-OPC1 cells for a total of 20 million cells; cohort dependent

SUMMARY:
The purpose of this study is to evaluate the safety of cross sequential escalating doses of AST-OPC1 administered among 5 cohorts at a single time-point between 21 and 42 days post injury, inclusively, to subjects with subacute cervical spinal cord injuries (SCI).

ELIGIBILITY:
Major Inclusion Criteria:

* Sensorimotor complete, traumatic SCI (ASIA Impairment Scale A) for cohorts 1,2,3
* Sensorimotor incomplete, traumatic SCI (ASIA Impairment Scale B) for cohorts 4,5
* Last fully preserved single neurological level (SNL) from C-4 to C-7
* From 18 through 69 years of age at time of injury
* Single spinal cord lesion on a post-stabilization magnetic resonance imaging (MRI) scan, with sufficient visualization of the spinal cord injury epicenter and lesion margins to enable post-injection safety monitoring
* Informed consent for this protocol and the companion long term follow-up protocol must be provided and documented (i.e., signed informed consent forms) no later than 37 days following injury
* Able to participate in an elective surgical procedure to inject AST-OPC1 21-42 days following SCI

Major Exclusion Criteria:

* SCI due to penetrating trauma
* Traumatic anatomical transection or laceration of the spinal cord based on prior surgery or MRI
* Any concomitant injury that interferes with the performance, interpretation or validity of neurological examinations
* Inability to communicate effectively with neurological examiner such that the validity of patient data could be compromised
* Significant organ damage or systemic disease that would create an unacceptable risk for surgery or immunosuppression
* History of any malignancy (except non-melanoma skin cancers)
* Pregnant or nursing women
* Body mass index (BMI) > 35 or weight > 300 lbs.
* Active participation in another experimental procedure/intervention

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward D Wirth III, MD, PhD, Study Director — Asterias Biotherapeutics
Locations (9):
- United States (9):
  - Univ. of California at San Diego, La Jolla, California
  - Rancho Los Amigos/USC, Los Angeles, California
  - Stanford University/Santa Clara Valley Medical Center, San Jose, California
  - Shepherd Center, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Thomas Jefferson University/Magee Rehabilitation, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fessler RG, Ehsanian R, Liu CY, Steinberg GK, Jones L, Lebkowski JS, Wirth ED, McKenna SL. A phase 1/2a dose-escalation study of oligodendrocyte progenitor cells in individuals with subacute cervical spinal cord injury. J Neurosurg Spine. 2022 Jul 8;37(6):812-820. doi: 10.3171/2022.5.SPINE22167. Print 2022 Dec 1. PMID 35901693
- [Derived] McKenna SL, Ehsanian R, Liu CY, Steinberg GK, Jones L, Lebkowski JS, Wirth E, Fessler RG. Ten-year safety of pluripotent stem cell transplantation in acute thoracic spinal cord injury. J Neurosurg Spine. 2022 Apr 1;37(3):321-330. doi: 10.3171/2021.12.SPINE21622. Print 2022 Sep 1. PMID 35364569

RESULTS

PARTICIPANT FLOW:
Groups:
- AST-OPC1, Cohort 1: n=3 subjects Dosage of 2 million cells AIS score A
- AST-OPC1, Cohort 2: n=6 subjects Dosage 10 million cells AIS score A
- AST-OPC1, Cohort 3: n=6 subjects Dosage of 20 million cells AIS score A
- AST-OPC1, Cohort 4: n=6 subjects Dosage of 10 million AIS score B
- AST-OPC1, Cohort 5: n=4 subjects Dosage of 20 million cells AIS score B
Period: Overall Study
Arm/Group | AST-OPC1, Cohort 1 | AST-OPC1, Cohort 2 | AST-OPC1, Cohort 3 | AST-OPC1, Cohort 4 | AST-OPC1, Cohort 5
Started | 3 | 6 | 6 | 6 | 4
Completed | 3 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics and demographic are described separately by each cohorts per Age, gender, race, height, weight, BMI
Groups:
- AST-OPC1, Cohort 1: n=3 Dosage of 2 million cells AIS score A
- AST-OPC1, Cohort 2: n=6 Dosage of 10 million cells AIS score A
- AST-OPC1, Cohort 3: n=6 Dosage of 20 million cells AIS score A
- AST-OPC1, Cohort 4: n=6 Dosage of 10 million cells AIS score B
- AST-OPC1, Cohort 5: n=4 Dosage of 20 million cells AIS score B
- Total: Total of all reporting groups
Arm/Group | AST-OPC1, Cohort 1 | AST-OPC1, Cohort 2 | AST-OPC1, Cohort 3 | AST-OPC1, Cohort 4 | AST-OPC1, Cohort 5 | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 4 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 6 | 6 | 4 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (6.1) | 24.5 (7.4) | 44.7 (14.7) | 28.5 (14.1) | 34.3 (20.7) | 30.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2 | 4
  Male | 3 | 5 | 5 | 6 | 2 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 3 | 5 | 6 | 6 | 2 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 6 | 6 | 4 | 25
The Abbreviated Injury Scale (AIS) [Count of Participants; unit: Participants] | 3 | 6 | 6 | 6 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Within 1 Year (365 Days) That Are Related to AST-OPC1 Injection
Description: Numbers of adverse events within 1 year (365 days) that are related to AST-OPC1 injection
Time Frame: One Year
Population: All 25 subject experienced at least one (1) AEs. The population description described on comment [1] above.
Measure: Number; unit: Adverse Events
Arm/Group | AST-OPC1, Cohort 1 | AST-OPC1, Cohort 2 | AST-OPC1, Cohort 3 | AST-OPC1, Cohort 4 | AST-OPC1, Cohort 5
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 4
Adverse Events | 92 | 122 | 133 | 118 | 69

2. Secondary Outcome: Neurological Function as Measured by Upper Extremity Motor Scores and Motor Level on International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examinations as Secondary End Point - 365 Days After Injection of AST-OPC1
Description: The scale is based on the ISNCSCI (International Standards for Neurological Classification of Spinal Cord Injury) that measures the severity of Spinal cord injury. The data was collected per time point during the first year (30,60,90,180,270,365). The 365-days time point was pre-specified as Secondary Outcome Measure. High score means better outcome. Units are "Scores on a scale".
  The score is divided to motor scale (0-100) and sensor scale (0-224).
  Motor scale is divided to subscale of upper extremity (0-50) and lower extremity (0-50).
  Upper and lower extremity are divided to subscale of Right (0-25) + Left (0-25).
  Each upper & lower extremity is divided to subscale of 5 motor nerve function (0-5).
  Sensor scale is divided to subscale of light touch (0-112) and pin prick (0-112).
  light touch and pin prick are divided to subscales of Right (0-56) + Left (0-56).
  Each right and left light touch and pin prick are divided to subscales of 28 sensor nerve function (0-2)
Time Frame: One Year
Measure: Mean (Full Range); unit: Score on a scale
Groups:
- AST-OPC1, Cohort 1: n=3 Dosage of 2 million AIS A
- AST-OPC1, Cohort 2: n=6 Dosage of 10 million AIS A
- AST-OPC1, Cohort 3: n=6 Dosage of 20 million AIS A
- AST-OPC1, Cohort 4: n=6 Dosage of 10 million AIS B
- AST-OPC1, Cohort 5: n=4 Dosage of 20 million AIS B
Arm/Group | AST-OPC1, Cohort 1 | AST-OPC1, Cohort 2 | AST-OPC1, Cohort 3 | AST-OPC1, Cohort 4 | AST-OPC1, Cohort 5
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 4
Score on a scale
  UEMS (Upper Extremities Motor Scale) - Baseline | 19 [0 to 50] | 21 [0 to 50] | 17 [0 to 50] | 22 [0 to 50] | 18 [0 to 50]
  UEMS (Upper Extremities Motor Scale) - Day 365 | 24 [0 to 50] | 34 [0 to 50] | 26 [0 to 50] | 28 [0 to 50] | 24 [0 to 50]
  LEMS (Lower Extremities Motor Scale) - Baseline | 0 [0 to 50] | 0 [0 to 50] | 0 [0 to 50] | 0 [0 to 50] | 0 [0 to 50]
  LEMS (Lower Extremities Motor Scale) - Day 365 | 0 [0 to 50] | 0 [0 to 50] | 0 [0 to 50] | 1 [0 to 50] | 1 [0 to 50]
  LT (Light Touch) - Baseline | 21 [0 to 112] | 27 [0 to 112] | 22 [0 to 112] | 35 [0 to 112] | 53 [0 to 112]
  LT (Light Touch) - Day 365 | 21 [0 to 112] | 32 [0 to 112] | 31 [0 to 112] | 46 [0 to 112] | 65 [0 to 112]
  PP (Pin Prick) - Baseline | 22 [0 to 112] | 23 [0 to 112] | 19 [0 to 112] | 25 [0 to 112] | 22 [0 to 112]
  PP (Pin Prick) - Day 365 | 20 [0 to 112] | 25 [0 to 112] | 21 [0 to 112] | 28 [0 to 112] | 34 [0 to 112]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | AST-OPC1, Cohort 1 | AST-OPC1, Cohort 2 | AST-OPC1, Cohort 3 | AST-OPC1, Cohort 4 | AST-OPC1, Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 4/6 | 2/6 | 1/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/6 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AST-OPC1, Cohort 1 (N=3) | AST-OPC1, Cohort 2 (N=6) | AST-OPC1, Cohort 3 (N=6) | AST-OPC1, Cohort 4 (N=6) | AST-OPC1, Cohort 5 (N=4)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered Mental Status (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspiration Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilateral Decubitus Ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilateral Hip Effusions (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilateral Pyelonephritis due to UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Buttock Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal Fluid Leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia Coli Urinary Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected Epidural Fluid (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Femoral Shaft Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Traumatic Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (UTI) (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02302157/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT02302157/SAP_001.pdf